CLINICAL TRIAL: NCT02920476
Title: A Phase II Trial of TAS-102 in Previously Treated Unresectable or Metastatic Squamous Cell Carcinoma of the Lung
Brief Title: TAS-102 in Previously Treated Unresectable or Metastatic Squamous Cell Lung Carcinoma (UF-STO-LUNG-003)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201601359 -A; UF-STO-LUNG-003 (Other: University of Florida); IIT-USA-0113 (Other: Taiho Oncology); OCR15277 (Other: University of Florida)
Record Dates: First submitted 2016-09-27; First posted 2016-09-30 (Estimated); Results first posted 2019-12-17 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-05

CONDITIONS: Squamous Cell Lung Carcinoma
Keywords: lung; metastatic; carcinoma
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): TAS-102
  Interventions: Drug: TAS-102

INTERVENTIONS:
Drug: TAS-102 — Days 1 through 5: TAS-102 (35 mg/m2/dose) orally 2 times daily with the first dose administered in the morning of Day 1 of each cycle and the last dose administered in the evening of Day 5. TAS-102 is to be taken within 1 hour of completion of morning and evening meals.
  Days 6 through 7: Rest
  Days 8 through 12: TAS-102 (35 mg/m2/dose) orally 2 times daily with the first dose administered in the morning of Day 8 of each cycle and the last dose administered in the evening of Day 12.
  Days 13 through 28: Rest
  Other Names: Lonsurf

SUMMARY:
This is a non-randomized, open label, sequentially enrolling phase II study with a Simon two-step enrollment design to evaluate the activity of TAS-102 in previously treated unresectable or metastatic squamous non-small cell cancer after progression through or intolerance to prior systemic therapy. The trial therapy of TAS-102 is to be administered orally at 35 mg/m2 each dose twice daily. The primary objective of the trial is to determine the progression-free survival, in months, of subjects receiving TAS 102 for the treatment of unresectable or metastatic recurrent squamous non-small cell lung cancers.

ELIGIBILITY:
Inclusion Criteria:

* Those who will be eligible will be all patients with unresectable and/or metastatic squamous cell non-small cell lung cancer who have disease which has been previously treated with an Food & Drug Administration (FDA)- or National Comprehensive Cancer Network (NCCN)-approved platinum doublet. Patients who have not received such therapy must have medical reasons for not receiving such therapy. Those who have a molecularly targetable genetic mutation in their tumor must have also received the appropriate specific therapy for that mutation. All will be appropriate candidates for chemotherapy treatment.

Subjects must meet all of the additional following criteria to be eligible for study participation:

* Eastern Cooperative Oncology Group (ECOG) Performance Status <2
* Life expectancy > 12 weeks
* Male or female' age >18 years
* Patients of childbearing potential must be using an effective means of contraception.
* Histologic diagnosis of squamous non-small cell lung cancer that has been treated adequately in the metastatic or unresectable setting with a platinum doublet chemotherapy regimen and now has evidence of disease progression. Patients may have also received additional chemotherapy, such as an immune checkpoint inhibitor or no more than one additional cytotoxic agent (thus participants may have received between one to three prior lines of therapy for metastatic or unresectable disease).
* Patients who have received platinum-based doublet therapy in the neoadjuvant or adjuvant setting will only be eligible if they have experienced disease progression after their last dose of cytotoxic chemotherapy.
* Patients who have a neoplasm for which there currently exists an FDA-approved targeted therapy (such as to epidermal growth factor receptor [EGFR] activating mutations, or ALK or ROS1 gene rearrangements) must have received all such targeted therapies and either exhibited progressive disease through such treatments, or have been shown to be intolerant of such therapies, prior to enrollment on this study.
* Baseline laboratory values (bone marrow, renal, hepatic):
* Adequate bone marrow function:
* Absolute neutrophil count >1000/µL
* Platelet count >100'000/µL
* Renal function:
* Serum creatinine < 2.0 mg/dL
* Hepatic function:
* Bilirubin <1.5x upper limit of normal (ULN)
* Serum calcium < 12 mg/dL
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for at least 6 months after the last dose of study drug to minimize the risk of pregnancy. Prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. WOCBP include any woman who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who is not post-menopausal. Post-menopause is defined as:
* Amenorrhea that has lasted for ≥ 12 consecutive months without another cause, or
* For women with irregular menstrual periods who are taking hormone replacement therapy (HRT), a documented serum follicle-stimulating hormone (FSH) level of greater than 35 mIU/mL.
* Males with female partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for 3 months following the last dose of study drug.
* Subjects must have provided written informed consent and be willing to comply with all study-related procedures.

Exclusion Criteria:

* Pregnant or lactating females
* Patients with a mixed histology NSCLC, such as adenosquamous carcinoma, where the squamous component is <50% of the assessed lesion
* Patients with a mixed histology where there are any small cell elements
* Patients who have not received and progressed through, refused, or been intolerant of, a commonly utilized platinum-doublet therapy (cisplatin or carboplatin paired with docetaxel, paclitaxel, nab-paclitaxel, gemcitabine, vinorelbine, etoposide or irinotecan) administered for the treatment of unresectable or metastatic lung cancer.
* Patients who have not received the appropriate prior targeted therapy for their lung cancer if eligible
* Any invasive malignancy treated within 3 years prior to Cycle 1, Day 1
* Myocardial infarction or ischemia within the 6 months before Cycle 1' Day 1
* Uncontrolled' clinically significant dysrhythmia, or prolonged QT segment
* Uncontrolled malignant disease in the central nervous system (previously treated disease is eligible, provided it has been radiographically stable for at least four weeks)
* Radiotherapy within the 2 weeks before Cycle 1, Day 1. If any radiation has been administered to the target lesion there must be evidence of growth by radiographic assessments or physical examination
* Major surgery within the 2 weeks before Cycle 1, Day 1
* Any co morbid condition that' in the view of the attending physician' renders the patient at high risk from treatment complications
* Subjects unwilling to use an acceptable method to avoid pregnancy for the entire study period and for at least 24 weeks after the last dose of study drug.
* History of any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician.
* Prisoners or subjects who are involuntarily incarcerated.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.
* Subjects demonstrating an inability to comply with the study and/or follow-up procedures.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2021-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennie Jones, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Cancer Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: TAS-102
  TAS-102: Days 1 through 5: TAS-102 (35 mg/m2/dose) orally 2 times daily with the first dose administered in the morning of Day 1 of each cycle and the last dose administered in the evening of Day 5. TAS-102 is to be taken within 1 hour of completion of morning and evening meals.
  Days 6 through 7: Rest
  Days 8 through 12: TAS-102 (35 mg/m2/dose) orally 2 times daily with the first dose administered in the morning of Day 8 of each cycle and the last dose administered in the evening of Day 12.
  Days 13 through 28: Rest
Period: Overall Study
Arm/Group | Treatment Arm
Started | 4
Completed | 3
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 4
Age, Continuous [Mean (Full Range); unit: years] | 66.5 [60 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: To determine the percentage of subjects who achieve an objective response by RECIST 1.1 criteria. ORR is defined as the number of participants who achieved either a partial or complete response by RECIST 1.1 criteria. By these criteria, Complete Response (CR) is defined as the disappearance of all target lesions and Partial Response (PR) is defined as a decrease of at least 30% in the sum of the longest diameter of the target lesions. Subjects must have received at least 2 cycles of therapy to be evaluable for this outcome measure.
Time Frame: 1 year
Population: Only 2 of the 4 subjects accrued to the study were evaluable for treatment response.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 2
Participants | 0

2. Secondary Outcome: Clinical Benefit Rate
Description: To determine the percentage of subjects who derive clinical benefit by RECIST 1.1 criteria. The clinical benefit rate is defined as the percentage of subjects who achieved either a complete or partial response or stable disease by RECIST 1.1 criteria. RECIST 1.1 criteria defines a partial response as a decrease of the sum of the largest diameter each target lesion by at least 30%. A complete response is defined as the disappearance of all target lesions (except lymph nodes, whose short axis must measure 10 mm or less). By RECIST 1.1 criteria, a subject is considered to have stable disease when the sum of the largest diameter of the target lesions has neither decreased enough to qualify as a partial response not increased enough to qualify as progressive disease.
Time Frame: 1 year
Population: Only 2 of the 4 participants accrued were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 2
Participants | 0

3. Secondary Outcome: Overall Survival (OS)
Description: To determine the overall survival in days
Time Frame: 1095 days
Measure: Mean (Full Range); unit: days
Arm/Group | Treatment Arm
Number analyzed (Participants) | 4
days | 449.25 [165 to 1095]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time that informed consent was signed until 28 days after the last dose of study treatment. During this time frame, adverse event data was collected at the time informed consent was signed, on days 1 and 15 of each treatment cycle, and 28 days after the last dose of study treatment at a minimum. The time period over which adverse event data was collected ranged from 165 to 1,095 days.
Description: Adverse events were assessed by the principal investigator, the treating sub-investigator, and/or the study coordinator at the time informed consent was signed, on days 1 and 15 of each treatment cycle, and 28 days after the last dose of study treatment at a minimum. Adverse events were assessed by physical examination, labs, and subject self-reports. The time period over which adverse event data was collected ranged from 165 to 1,095 days.
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 4/4
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=4)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1
Respiratory infection (Infections and infestations) | 1
Non-cardiac chest pain (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=4)
Non-cardiac chest pain (General disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Dysgeusia (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Fatigue (General disorders) | 2
Fever (General disorders) | 1
Hot flashes (Vascular disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Neutrophil count decreased (Investigations) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 — shoulder pain
Platelet count decreased (Investigations) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Tremor (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/76/NCT02920476/Prot_SAP_000.pdf